CLINICAL TRIAL: NCT04579107
Title: KARMA Kontrast - a Controlled Clinical Trial Evaluating Contrast Enhanced Mammography in Early Detection of Breast Cancer
Brief Title: KARMA Kontrast Evaluating Contrast Enhanced Mammography in Early Detection of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Per Hall, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KARMA Kontrast
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Contrast Enhanced Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: The added Contrast Enhanced Mammography will be evaluated by a radiologist blinded from the radiologists evaluating the standard of care examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast Enhanced Mammography (Other): All included women go through a Contrast Enhanced Mammography added to the standard of care examinations.
  Interventions: Combination Product: Contrast Enhanced Mammography

INTERVENTIONS:
Combination Product: Contrast Enhanced Mammography — A modality for examining breast conditions which is already approved and used but the evaluation of its role in a recalled screening population is limited. Intravenous iodine contrast is given prior to the mammogram.

SUMMARY:
Women taking part in the National Mammography Screening Program, examined at Södersjukhuset Breast Centre at Södra station in Stockholm and recalled because of suspicion of breast cancer will be invited to participate. A Contrast Enhanced Mammography will be added to the standard of care procedures for investigating a suspicion of breast cancer and blinded from each other 2 radiologists will evaluate either the Contrast Enhanced Mammography or the standard of care examinations. When comparing the potentially extra findings with Contrast Enhanced Mammography will be calculated. Potential side effects together with the patient experience will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: >25 - <85 years
* Recalled after Mx screening based on abnormal mammographic findings or refered for breast cancer related symtoms
* The woman has read, understood and signed the Informed Consent Form (ICF)

Exclusion Criteria:

* Previous breast cancer
* A breast biopsy performed within 6 weeks preceding the study
* Recent exposure (during the last week) to iodine contrast media.
* Pregnancy
* Current breast feeding
* Diagnosed with a pheochromocytoma or a paraganglioma
* Diagnosed with myeloma or other malignant plasma cell disease
* Diagnosed with myasthenia gravis
* A renal failure or kidney disorder with increased risk for developing renal failure (single kidney or kidney transplanted)
* Diabetes (other than dietary treated)
* Heart failure or liver failure
* Intake of potentially nephrotoxic substances (daily intake of NSAID, nephrotoxic antibiotics or nephrotoxic chemotherapy)
* Iodine contrast allergy
* Uncontrolled thyrotoxicosis
* A history of severe allergy
* Subjects unable to read, understand and execute written informed consent
* Any medical aspect that, according to the investigator, could jeopardize the health of the participant

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Contrast Enhanced Mammography | 1 day
  Evaluating sensitivity of Contrast Enhanced Mammography in detecting multifocality and/or contralateral breast cancer, compared to standard breast radiology work-up methods.

SECONDARY OUTCOMES:
Specificity of Contrast Enhanced Mammography | 1 day
  Estimate the specificity of Contrast Enhanced Mammography in detecting absence of breast cancer, compared to standard breast radiology work-up methods.
Safety of Contrast Enhanced Mammography | 30 days
  Evaluate the safety of using Contrast Enhanced Mammography, based on adverse event reporting. Potential adverse event will be collected, reported and, if necessary, intervened, on the day for the Contrast Enhanced Mammography and up to 30 days after. All adverse events will be put in to the eCRF.
Patient acceptance of Contrast Enhanced Mammography | 30 days
  Evaluate the acceptance in patients, based on a questionnaire at the end of the study visit and structured telephone interviews 1-2 weeks after. The answers to the questionnaire is on a 5-grade scale. The interviews will go deeper and summaries of the answers will be put in to the eCRF.
Tumor size assessment | 1 day
  Comparing Contrast Enhanced Mammography with each standard breast radiology work-up method for tumor size assessment.
Mammographic density influence on the performance of Contrast Enhanced Mammography | 1 day
  Evaluate if mammographic density influences the performance of Contrast Enhanced Mammography compared to standard breast radiology work-up methods.
Contrast Enhanced Mammography costs | 1 day
  Calculate the costs for using Contrast Enhanced Mammography

CONTACTS AND LOCATIONS:
Overall Officials: Per Hall, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Bröstcentrum, Södersjukhuset, Stockholm, Sweden

REFERENCES:
- See also: Research group web page — https://karmastudy.org/